CLINICAL TRIAL: NCT01711398
Title: A Non-randomized, Open-label, Multi-centric Dose-finding Adaptive Phase I/IIa Study to Assess Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Repeated Intravenous IPP-204106N Administrations in Adult Patients With Advanced Solid Tumors
Brief Title: Dose-finding Adaptive Phase I/IIa Study to Assess Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of IPP-204106N on Advanced Solid Tumors
Acronym: IP N02
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elro Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP N02
Record Dates: First submitted 2012-10-09; First posted 2012-10-22 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: All Solid Tumors
Keywords: solid tumor; peptide
MeSH Terms: interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IPP204106N (Experimental)
  Interventions: Drug: Drug

INTERVENTIONS:
Drug: Drug

SUMMARY:
The experimental plan will consist in:

The dose-finding Bayesian adaptive phase I portion of the study is designed to determine the optimal and recommended dose of IPP-204106N using a Bayesian "with memory" design with combined toxicity and pharmacokinetic endpoints to determine doses for successive cohorts of three patients. The Bayesian methodology allows updating information as the trial progresses and stopping the trial as soon as the information obtained is deemed to be sufficient. Preclinical toxicokinetic studies of N6L and IPP-204106N in dogs and the first phase I clinical trial with N6L will be used to inform the prior distribution in the present study.

The decisional part, according to the results of the phase I portion of the study, will define the optimal dose recommended for the phase IIa portion of the study.

The phase IIa portion of the study will confirm the optimal dose, and is designed to evaluate the safety and the preliminary efficacy of IPP-204106N in an expanded patient population treated at the recommended dose of IPP-204106N.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to initiation of any study-specific procedures for study participation and signed informed consent for tumor biopsy. Informed consent for tumor biopsy is mandatory for patients included in the phase IIa part of the study.
* Man or woman at least 18 years of age.
* Histological or cytological confirmed advanced solid tumor, non eligible for curative local treatment or active palliation with systemic therapy.
* Patients with measurable or evaluable disease (by tumor measurements or by tumor biomarker) with a proof of disease progression. At least one measurable lesion is mandatory for the phase IIa portion of the study.
* Patients currently under treatment with N6L or patients who have taken part in the Phase I part of the study are eligible for the phase IIa part, according to the investigator's judgment, irrespective of their tumor status.
* Tumor biopsy available at study entry for patients included in the phase IIa part of the study and if possible for phase I patients.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Life expectancy more than 3 months according to the investigator's judgment.
* Recovery from any acute toxicity related to prior therapy. Toxicity should be ≤grade 1 according to NCI-CTCAE criteria or returned to baseline excluding alopecia.
* Adequate hematological counts: neutrophils >=1.5 x 109/L, platelets >=100 x 109/L, hemoglobin >=9 g/dL.
* Adequate renal function: serum creatinine ≤1.5 × upper limit of normal range (ULN).
* Adequate hepatic function:

  * Serum bilirubin ≤1.5 × ULN (except for isolated hyperbilirubinemia attributed to Gilbert's syndrome).
  * Alkaline phosphatase, aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT) ≤2.5 × ULN (or ≤5 × ULN in case of liver metastases).
* All women of child-bearing potential must use adequate contraception throughout the duration of the study, or their partner must be surgically sterilized. The pre-study pregnancy test must be negative for women with reproductive potential. Women who have been surgically sterilized or are at least two years post-menopausal may be enrolled and do not need birth control.

Exclusion Criteria:

* Hematological malignancy (including lymphomas).
* Any of the following within the 6 months prior to study drug administration: severe/unstable angina, myocardial infarction, coronary artery bypass graft, symptomatic congestive heart failure, stroke, including transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac arrhythmias of NCI-CTCAE grade ≥2.
* Active uncontrolled infections.
* Uncontrolled hypertension.
* Radiotherapy or chemotherapy within 4 weeks before study entry (6 weeks for nitrosoureas or mitomycin).
* Pregnancy or breastfeeding.
* Participation to another therapeutic clinical trial within the last 4 weeks except studies including treatment with N6L.
* History of severe allergic reactions.
* Documented or suspected allergy to any nucleolin antagonist.
* Documented allergy to excipient (mannitol or chondroitin sulfate) product.
* Documented allergy to aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Recommended optimal dose of intravenous IPP-204106N administered for at least 5 consecutive days. | up to 18 months
  Toxicity assessed during cycle 1 (until day 12): number of patients experiencing a dose limiting toxicity (DLT) according to the NCI-CTCAE (v 4.0, May 2009), defined as:
  * Hematological drug-related toxicity: grade 4 neutropenia ≥7 days, grade 4 thrombocytopenia, grade 3 thrombocytopenia with hemorrhage/bleeding, and febrile neutropenia.
  * Nausea, vomiting or diarrhea grade ≥3 despite optimal treatment.
  * Any other drug-related biological or clinical grade ≥3 toxicity.
  Plasma exposure assessed during cycle 1 (on day 1): number of patients reaching targeted plasma drug exposure, i.e. plasma N6L concentration ≥5 µM for at least two hours. This concentration corresponds to active concentration in vitro in human tumor cell lines.

SECONDARY OUTCOMES:
Overall safety of IPP-204106N. | up to 18 months
  number of participants with DLT
tumor response rate | up to 24 months
  Each patient's best objective response will be determined. The categories for best objective response are CR, PR, SD, PD or NE.
Time to progression (TTP) of IPP-204106N at the recommended dose. | up to 15 months
  Analysis of time to progression (TTP) will be performed using in the ITT population using non-parametric method of Kaplan Meier and survival curves (PROC LIFETEST with SAS® software).
genomic and proteomic tumor biomarkers identification | up to 15 months
  Genomic and/or proteomic biomarkers analyses may be performed as exploratory analyses, to identify the patients who, based on their individual tumor signature, will be most likely to respond and benefit from IPP-204106N therapy, and will be detailed in a further statistical analysis plan.
tumor response duration of objective responses | up to 15 months
  The duration of overall response is measured from the time measurement criteria are first met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study).
tumor response duration of stabilizations. | up to 15 months
  Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest summon study (if the baseline sum is the smallest, this is the reference for calculation of PD).
Progression-free survival (PFS) of IPP-204106N at the recommended dose. | up to 15 months
  Analysis of progression-free survival (PFS) will be performed using in the ITT population using non-parametric method of Kaplan Meier and survival curves.
To determine the pharmacokinetic (PK) profile of IPP-204106N during the dose-escalation phase of the study. | up to 18 months
to evaluate the tumor growth rate (GR) | up to 24 months
  The tumor GR analyses may be performed as exploratory analyses
To evaluate the early metabolic effects of IPP-204106N as measured by 18FDG-PET CT | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Isambert, Dr, Principal Investigator — Centre Georges Francois Leclerc
Locations (3):
- Institut Jules Bordet, Brussels, Belgium
- France (2):
  - Centre Georges François Leclerc, Dijon
  - Centre Claudius Regaud, Toulouse